CLINICAL TRIAL: NCT07268157
Title: Evaluation of the Effects of Computer-Controlled and Traditional Local Anesthesia on Pain and Anxiety in Children With Molar Incisor Hypomineralization
Brief Title: Evaluation of Different Anesthesias in Children With Molar Incisor Hypomineralization
Status: Completed | Type: Observational
Sponsor: Canan Bayraktar Nahir (Other)
Responsible Party: Sponsor-Investigator, Canan Bayraktar Nahir, Associate Professor, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Other Study IDs: 23-KAEK-205
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Molar-Incisor Hypomineralization
Keywords: Pain; Anxiety; Computer-Controlled Local Anesthesia; Molar Incisor Hypomineralization; Pediatric Dentistry
MeSH Terms: conditions — Molar Hypomineralization; Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maxilla: maxillary 1st molar
  Interventions: Device: Computer-controlled anesthesia device (SleeperOne); Procedure: Conventional injection technique
- Mandible: mandibular 1st molar
  Interventions: Device: Computer-controlled anesthesia device (SleeperOne); Procedure: Conventional injection technique

INTERVENTIONS:
Device: Computer-controlled anesthesia device (SleeperOne) — Intraosseous anesthesia administered with the computer-controlled anesthesia device (SleeperOne)
Procedure: Conventional injection technique — Anesthesia administered using the conventional injection technique

SUMMARY:
In children with molar-incisor hypomineralization (MIH), insufficient depth of anesthesia can lead to increased anxiety and behavior management problems, which may negatively affect the quality of restorations. This situation has increased the need for modern techniques and devices to minimize pain during local anesthesia. The aim of this study was to compare the effects of the SleeperOne computer-controlled local anesthesia system and the conventional local anesthesia technique on pain and anxiety in children with MIH. The null hypothesis of the study stated that there would be no statistically significant difference between the effects of the two local anesthesia methods on pain and anxiety in children with MIH.

DETAILED DESCRIPTION:
The study was conducted using a split-mouth design with 28 patients and 56 teeth who met the inclusion criteria and were recruited from the Department of Pediatric Dentistry, Faculty of Dentistry, Tokat Gaziosmanpaşa University. The patients included in the study were randomly assigned to two groups:

* Control group: Anesthesia administered using the conventional injection technique.
* Study group: Intraosseous anesthesia administered with the computer-controlled anesthesia device (SleeperOne).

Teeth affected by MIH were classified according to the Molar-Incisor Hypomineralization Treatment Need Index (MIH-TNI). Those in category 2 were evaluated as "Without hypersensitivity," while those in category 4 were assessed as "With hypersensitivity" Prior to the study, all participants completed the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS). Pulse rate, oxygen saturation (SpO₂), and salivary cortisol levels were measured before local anesthesia, after anesthesia, and after treatment. In addition, the Wong-Baker FACES Pain Rating Scale (WBS), Visual Analogue Scale (VAS), and Face, Legs, Activity, Cry, Consolability Scale (FLACC) were used. The data were analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 6 and 12
* Not having a systemic disease
* Frankl Behavior Rating Scale score of 3 or 4
* Presence of bilateral MIH in the lower or upper jaw permanent first molars
* Deep dentinal caries in permanent 1st molars that can be treated with vital pulp treatments
* No history of acute pain in the teeth planned to be included in the study

Exclusion Criteria:

* Having a systemic disease
* Allergy to the anesthetic to be used
* Having an acute infection
* Unilateral teeth with BAKH lesions and deep dentin caries
* If they or their parents do not want to participate in the study
* The teeth planned to be included in the study showed irreversible pulpitis symptoms
* Among the patients planned to be included in the study; those who did not consent to anesthesia or treatment, those who did not come to their second appointment, and those who needed devital pulp treatments during the procedure

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 6-12 years old who apply to Tokat Gaziosmanpaşa University, Faculty of Dentistry, Department of Pedodontics.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of different anesthesia on pain in teeth with MIH | 6 month
  VAS (Visual Analog Scale), WBS (Wong-Baker Facial Rating Scale for Pain) and FLACC (Face, Leg, Activity, Crying, Consolability Behavioral Pain Rating Scale) scales were used for pain assessment. In the VAS, patients were asked to select the number expressing the level of pain from a linear scale with numerical values between 0-10 (0 no pain, 10 excruciating pain). On the WBS scale, they were asked to choose one of six faces, with the happy face at 0 symbolizing "no pain" and the crying face at 5 symbolizing "the most pain". Both numerical (VAS) and visual (WBS) assessments were made. According to the scores obtained on the FLACC scale: 0 points indicated that the patient was relaxed and peaceful, 1 to 3 points indicated mild discomfort, 4 to 6 points indicated moderate pain and 7 to 10 points indicated severe pain.
Evaluation of the effect of different anesthesia on anxiety in teeth with MIH | 6 month
  The Child Fear Rating Scale-Dental Subscale (CFSS-DS), a numerical scale, was used to assess anxiety in patients. According to the answers given in the CFSS-DS; a score between 15 and 75 is obtained. According to the score; it was accepted that children aged 15-38 years did not have dental anxiety, while children with a score of 38 and above were considered to have dental anxiety.
  Pulse rate, oxygen saturation and salivary cortisol measurements were used in an anxiety assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanapaş University, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
with the link to be prepared later

REFERENCES:
- [Result] Smail-Faugeron V, Muller-Bolla M, Sixou JL, Courson F. Evaluation of intraosseous computerized injection system (QuickSleeper) vs conventional infiltration anaesthesia in paediatric oral health care: A multicentre, single-blind, combined split-mouth and parallel-arm randomized controlled trial. Int J Paediatr Dent. 2019 Sep;29(5):573-584. doi: 10.1111/ipd.12494. Epub 2019 Apr 8. PMID 30883951
- See also: Evaluation of intraosseous computerized injection system (QuickSleeper™) vs conventional infiltration anaesthesia in paediatric oral health care: A multicentre, single-blind, combined split-mouth and parallel-arm randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/30883951/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT07268157/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT07268157/ICF_001.pdf